CLINICAL TRIAL: NCT00238160
Title: Phase III Randomized Study of Surgical Resection With Versus Without Postoperative Hepatic Arterial Chemotherapy in Patients With Hepatocellular Carcinoma and Portal Vein Tumor Thrombus
Brief Title: Surgery With or Without Hepatic Arterial Chemotherapy in Treating Patients With Liver Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Kyoto University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: KYUH-UHA-HCC02-01; CDR0000363800 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-10-12; First posted 2005-10-13 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2006-07

CONDITIONS: Localized Resectable Adult Primary Liver Cancer; Stage III Childhood Liver Cancer
MeSH Terms: interventions — Cisplatin; Fluorouracil; Chemotherapy, Adjuvant; Drug Therapy; Surgical Procedures, Operative

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: adjuvant therapy
Procedure: chemotherapy
Procedure: conventional surgery
Procedure: hepatic arterial infusion
Procedure: surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving drugs directly into the arteries around the tumor may kill more tumor cells. Giving chemotherapy after surgery may kill any remaining tumor cells. It is not yet known whether surgery and hepatic arterial chemotherapy are more effective than surgery alone in treating patients with liver cancer that has spread to the portal vein.

PURPOSE: This randomized phase III trial is studying surgery and hepatic arterial chemotherapy to see how well they work compared to surgery alone in treating patients with liver cancer that has spread to the portal vein.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of surgical resection with vs without postoperative hepatic arterial chemotherapy in patients with hepatocellular carcinoma and portal vein tumor thrombus.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to grade of portal invasion and Child-Pugh classification. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo macroscopic curative resection. Within 28 days after surgery, patients without post-surgery complications undergo hepatic arterial infusion comprising fluorouracil and cisplatin on days 1-5, 8-12, and 15-19. Treatment continues for 6 months.
* Arm II: Patients undergo macroscopic curative resection.

PROJECTED ACCRUAL: A total of 100 patients (50 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed hepatocellular carcinoma (HCC) with portal vein tumor thrombus
* Tumor thrombus in the main trunk or first branch of the portal vein
* No apparent distant metastases on chest CT scan and bone scintigraphy within the past 6 weeks
* No pleural effusion or ascites

PATIENT CHARACTERISTICS:

Age

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Neutrophil count > 1,000/mm^3
* Platelet count > 50,000/mm^3
* Hemoglobin > 8 g/dL

Hepatic

* Bilirubin < 2 times upper limit of normal (ULN)
* ALT and AST < 4 times ULN

Renal

* Creatinine normal

Cardiovascular

* No severe heart disease
* No cardiac effusion

Other

* No other malignant disease
* No high risk for esophageal varices rupture
* No allergy to fluorouracil or cisplatin

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior hepatic arterial chemotherapy
* No prior systemic chemotherapy for HCC

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Iwao Ikai, MD, Study Chair — Kyoto University Hospital
Locations (4):
- Japan (4):
  - Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto City Hospital, Kyoto
  - Kyoto University Hospital, Kyoto
  - Kyoto-Katsura Hospital, Kyoto